CLINICAL TRIAL: NCT03032653
Title: Immediate Unprotected Weight-Bearing and Range of Motion After Open Reduction and Internal Fixation of Unstable Ankle Fractures. A Historical Control Group Comparative Study
Brief Title: Immediate Weight-Bearing Ankle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHREB #: 2016-101
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Ankle Fractures; Surgery
Keywords: ankle, fracture, rehabilitation, weightbearing, early, late
MeSH Terms: conditions — Ankle Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late WB (Active Comparator): Intervention: Patients receive a plaster splint in the operating room. They are not permitted to WB or ROM on the affected limb at this stage. At the first follow-up appointment (two weeks post-op), the splint is removed and a removable pre-fabricated walking boot applied. At this stage the patient is permitted to WB as tolerated while wearing the boot, and to perform ROM exercises with the boot removed. At six weeks post-op, the boot is discontinued and full unrestricted and unprotected weightbearing and ROM is permitted.
  Interventions: Other: Late Rehabilitation
- Immediate unprotected WB and ROM (Experimental): Patient do NOT receive a brace or splint of any kind. They are permitted to weightbear and range of motion as tolerated within the limitations of their own comfort. Use of ambulatory aids of any kind is permitted as needed without restrictions.
  Interventions: Other: Early Rehabilitation

INTERVENTIONS:
Other: Late Rehabilitation — Post-0p: Non weight-bearing and no range of motion for 2 weeks post treatment. 2 weeks: Splint removed, removable pre-fabricated walking boot applied. WB as tolerated with boot, range of motion out of boot.
  6 weeks: Boot discontinued and full unrestricted and unprotected WB and ROM permitted 6 weeks:
  Arms: Late WB
Other: Early Rehabilitation — Weightbearing and range of motion as tolerated within the limitations of participant's own comfort. Use of ambulatory aides of any kind is permitted as needed without restriction. No brace or splint of any kind is permitted
  Arms: Immediate unprotected WB and ROM

SUMMARY:
This single-centre historical control group comparative study will compare outcomes of surgically-treated rotational ankle fractures and the current routine practice of early protected weightbearing and range of motion with immediate unprotected weightbearing as tolerated and range of motion after ankle open reduction and internal fixation.

DETAILED DESCRIPTION:
Ankle fractures are among the most common injuries, making up 9% of all fractures. Rotational ankle fractures are among the most common of all fractures, with an incidence averaging 4.2 per 1,000 individuals annually. These fractures range from minimal injuries amenable to non-surgical management to complex injuries with potential of long-term sequelae. Known risk factors for ankle fractures are age, body mass index and previous ankle fracture, with the highest incidence in elderly women.

Most ankle fractures are low-energy injuries which occur when the body rotates about a planted foot, whether it be during sports, normal gait, or otherwise. Stable ankle fractures are generally treated non-surgically, while unstable fractures are usually treated with surgical reduction and fixation, with indications previously well-described and published.

However, the post-operative management of such injuries is still controversial, with large variability between care providers. Protocols range from complete immobilization of the affected ankle and non-weightbearing to early range-of-motion (ROM) and weightbearing (WB). Studies have compared immobilization and non-WB to early ROM and WB but results have been mixed, with the most recent study demonstrating safety and advantages to protected WB and ROM at two weeks post-operatively versus non-WB and immobilization for six weeks.

The Investigators intend to expand on the studies above and propose a single-centre historical control group comparative study to compare outcomes of surgically-treated rotational ankle fractures and the current routine practice of early protected weightbearing and range of motion with immediate unprotected weightbearing as tolerated and range of motion after ankle open reduction and internal fixation.

ELIGIBILITY:
Inclusion Criteria:

* lateral malleolus fracture with talar shaft
* vertical shear medial malleolus fracture without superior articular involvement
* bimalleolar fracture
* any ankle fracture with posterior malleolus fragment involving 25% or less of the articular surface on the lateral ankle radiograph
* 43.B1 (pure split of distal tibia - but only if does not involve any of tibial plafond, i.e., only the vertical split of medial malleolus)
* 44.A1 (Weber A)
* 44.A2 (Bimalleolar)
* 44.A3 (posterior malleolus involvement - but only if < 25% articular involvement on lateral x-ray)
* 44-B1 (Isolated)
* 44.B2 (with medial lesion)
* 44.B3 (with medial lesion & Volkmann's #)
* closed, Gustilo-Anderson Grade I or Grade II open fractures are included
* willing and able to sign the consent
* willing and able to follow the protocol and attend follow-up visits
* able to read and understand English or have an interpreter available

Exclusion Criteria:

* skeletal immaturity demonstrated radiographically by open physes
* previous ipsilateral ankle surgery
* bilateral ankle fractures
* non ambulatory prior to injury
* inability to comply with postoperative protocol (i.e., cognitive impairment)
* medical comorbidity precluding surgery
* poorly controlled diabetes (i.e. dense neuropathy / hx of ulcers / sensory deficit)
* polytrauma patients (other injuries involving the ipsi/contralateral lower limbs, including the hip, that would interfere with mobilization/rehabilitation)
* surgical date > 14 days (time of injury to OR)
* Gustilo-Anderson grade III open fractures
* tibial plafond fractures
* active infection at the surgical site diagnosed clinically by the attending surgeon
* any ankle fracture with posterior malleolus fragment involving more than 25% of the articular surface on the lateral ankle radiograph
* any medial malleolus fracture involving the superior articular surface
* any ankle fracture requiring syndesmosis fixation
* any ankle fracture-dislocation
* incarceration
* likely problems, in the judgment of the investigator, with maintaining follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Olerud and Molander Score | 6 weeks post treatment
  An assessment of symptoms after ankle fracture.

SECONDARY OUTCOMES:
EQ-5D | 2, 6 and 12 weeks post treatment
  Health Related quality of life outcome measure using five dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
WPAI:SHP Work Productivity and Activity Impairment Questionnaire: Specific Health Problem | 2, 6 and 12 weeks post treatment
  A questionnaire pertaining to the effect of the participant's ankle fracture on their ability to work and perform regular activities.
Range of Motion | 2, 6 and 12 weeks post treatment
  Amount of ankle dorsiflexion and plantarflexion (measured in degrees) as determined by goniometer assessment, as well as total arc of ankle ROM (dorsiflexion+ plantarflexion). This will be measured on both ankles for comparison.
Wound Healing | 2, 6 and 12 weeks post treatment
  Complications regarding the surgical wound, including but not limited to signs of infection or dehiscence.
Fracture Healing | 2, 6 and 12 weeks post treatment
  Radiographic assessment to determine healing, loss of reduction, loss of hardware fixation, or ankle alignment.
Need for Re-operation | 2, 6 and 12 weeks post treatment
  Any issue, whether it be a wound complication or fracture complication, requiring re-operation.
Time to Return to Work | 2, 6 and 12 weeks post treatment
  The chronological time between the date of surgery to the first day the participant returned to occupational duties, if currently employed and returns to work within the 12 weeks postoperative follow-up period. For the purposes of this study, students enrolled in educational activities will have their schooling treated as their occupational duty.
Radiographic assessment | 2, 6 and 12 weeks post treatment
  Assessment of alignment, hardware fixation, fracture reduction and loss of reduction (defined as any shft of 2mm or more in fracture position)

CONTACTS AND LOCATIONS:
Overall Officials: Darius G Viskontas, MD, FRCSC, Principal Investigator — Royal Columbian Hospital / Fraser Health Authority; Vu (Brian) Le, MD, FRSCS, Principal Investigator — Royal Columbian Hospital / Fraser Health Authority; Kelly L Apostle, MD, FRCSC, Principal Investigator — Royal Columbian Hospital / Fraser Health Authority
Locations (1):
- Royal Columbian Hospital / Fraser Health Authority, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Hoelsbrekken SE, Kaul-Jensen K, Morch T, Vika H, Clementsen T, Paulsrud O, Petursson G, Stiris M, Stromsoe K. Nonoperative treatment of the medial malleolus in bimalleolar and trimalleolar ankle fractures: a randomized controlled trial. J Orthop Trauma. 2013 Nov;27(11):633-7. doi: 10.1097/BOT.0b013e31828e1bb7. PMID 23454858
- [Background] Petrisor BA, Poolman R, Koval K, Tornetta P 3rd, Bhandari M; Evidence-Based Orthopaedic Trauma Working Group. Management of displaced ankle fractures. J Orthop Trauma. 2006 Jul;20(7):515-8. doi: 10.1097/00005131-200608000-00012. PMID 16891946
- [Background] Michelson JD, Magid D, McHale K. Clinical utility of a stability-based ankle fracture classification system. J Orthop Trauma. 2007 May;21(5):307-15. doi: 10.1097/BOT.0b013e318059aea3. PMID 17485995
- [Background] Dehghan N, McKee MD, Jenkinson RJ, Schemitsch EH, Stas V, Nauth A, Hall JA, Stephen DJ, Kreder HJ. Early Weightbearing and Range of Motion Versus Non-Weightbearing and Immobilization After Open Reduction and Internal Fixation of Unstable Ankle Fractures: A Randomized Controlled Trial. J Orthop Trauma. 2016 Jul;30(7):345-52. doi: 10.1097/BOT.0000000000000572. PMID 27045369
- [Background] Gul A, Batra S, Mehmood S, Gillham N. Immediate unprotected weight-bearing of operatively treated ankle fractures. Acta Orthop Belg. 2007 Jun;73(3):360-5. PMID 17715727
- [Background] O'Sullivan ME, Bronk JT, Chao EY, Kelly PJ. Experimental study of the effect of weight bearing on fracture healing in the canine tibia. Clin Orthop Relat Res. 1994 May;(302):273-83. PMID 8168314
- [Background] Lehtonen H, Jarvinen TL, Honkonen S, Nyman M, Vihtonen K, Jarvinen M. Use of a cast compared with a functional ankle brace after operative treatment of an ankle fracture. A prospective, randomized study. J Bone Joint Surg Am. 2003 Feb;85(2):205-11. doi: 10.2106/00004623-200302000-00004. PMID 12571295
- [Background] Honigmann P, Goldhahn S, Rosenkranz J, Audige L, Geissmann D, Babst R. Aftertreatment of malleolar fractures following ORIF -- functional compared to protected functional in a vacuum-stabilized orthesis: a randomized controlled trial. Arch Orthop Trauma Surg. 2007 Apr;127(3):195-203. doi: 10.1007/s00402-006-0255-x. Epub 2006 Dec 30. PMID 17195934
- [Background] van Laarhoven CJ, Meeuwis JD, van der WerkenC. Postoperative treatment of internally fixed ankle fractures: a prospective randomised study. J Bone Joint Surg Br. 1996 May;78(3):395-9. PMID 8636173
- [Background] Ahl T, Dalen N, Lundberg A, Bylund C. Early mobilization of operated on ankle fractures. Prospective, controlled study of 40 bimalleolar cases. Acta Orthop Scand. 1993 Feb;64(1):95-9. doi: 10.3109/17453679308994541. PMID 8451961
- [Background] Finsen V, Saetermo R, Kibsgaard L, Farran K, Engebretsen L, Bolz KD, Benum P. Early postoperative weight-bearing and muscle activity in patients who have a fracture of the ankle. J Bone Joint Surg Am. 1989 Jan;71(1):23-7. PMID 2492286
- [Background] Cimino W, Ichtertz D, Slabaugh P. Early mobilization of ankle fractures after open reduction and internal fixation. Clin Orthop Relat Res. 1991 Jun;(267):152-6. PMID 2044269
- [Background] Hedstrom M, Ahl T, Dalen N. Early postoperative ankle exercise. A study of postoperative lateral malleolar fractures. Clin Orthop Relat Res. 1994 Mar;(300):193-6. PMID 8131334
- [Background] Egol KA, Dolan R, Koval KJ. Functional outcome of surgery for fractures of the ankle. A prospective, randomised comparison of management in a cast or a functional brace. J Bone Joint Surg Br. 2000 Mar;82(2):246-9. PMID 10755435
- [Background] Smeeing DP, Houwert RM, Briet JP, Kelder JC, Segers MJ, Verleisdonk EJ, Leenen LP, Hietbrink F. Weight-bearing and mobilization in the postoperative care of ankle fractures: a systematic review and meta-analysis of randomized controlled trials and cohort studies. PLoS One. 2015 Feb 19;10(2):e0118320. doi: 10.1371/journal.pone.0118320. eCollection 2015. PMID 25695796